CLINICAL TRIAL: NCT02815956
Title: InteresT And Mechanisms of Percutaneous Posterior tIbial Nerve Stimulation to Prevent pOstoperative Ileus in ColorectAl Surgery: A Preliminary Study
Brief Title: Tibial Nerve Stimulation and Postoperative Ileus
Acronym: pre-TAPIOCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-A00438-43
Record Dates: First submitted 2016-06-16; First posted 2016-06-28 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Postoperative Ileus
Keywords: percutaneous tibial nerve stimulation; randomized; controlled study

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- percutaneous tibial nerve stimulation (ST) (Experimental): Stimulation the day before surgery (x1), 30 minutes Stimulation the day of surgery, before surgery (at least 2 hours before surgery) and after surgery.
  Stimulation every day (x3) after surgery until gastrointestinal functions recovery.
  The protocol of stimulation is the same, that the one performed for fecal incontinence.
  Interventions: Device: percutaneous tibial nerve stimulation
- placebo (P) (Placebo Comparator): Stimulation the day before surgery (x1), 30 minutes Stimulation the day of surgery, before surgery (at least 2 hours before surgery) and after surgery.
  Stimulation every day (x3) after surgery until gastrointestinal functions recovery.
  The device delivers ineffective impulses.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: percutaneous tibial nerve stimulation
  Arms: percutaneous tibial nerve stimulation (ST)
Device: Placebo
  Arms: placebo (P)

SUMMARY:
Postoperative ileus (POI) causes patient's discomfort and leads to an increase of cost of management after colorectal surgery because of an increase of the morbidity rate or of the rate of early rehospitalization after discharge.

Enhanced recovery programs allowed a reduction of its rate but 20 to 30% of patients will experiment POI.

A new approach during preoperative era, using mastication or preoperative physical activity, has been proposed to improve postoperative course. This leads to a vagal activation (action especially on upper GI).

Sacral stimulation using percutaneous tibial nerve stimulation (PTNS) has an effect on lower GI.

The aim of this study was to assess the efficacy and the feasibility of PTNS during perioperative course, to prevent POI with respect with placebo.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years
* elective colectomy or proctectomy
* agreement for the research

Exclusion Criteria:

* chronic inflammatory bowel disease
* irritable bowel disease documented
* history of surgery on oesophagus or stomach
* acetylcholine dysfunction
* enterostoma
* patient holder of pace-maker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06-09 (Actual)

PRIMARY OUTCOMES:
delay before solid food tolerance and first stool recovery (expressed in days afters surgery). Day 0 (D0) is the day of surgery. | data collected from 6 hours after the end of surgery to the recovery. This recovery is expected to be between 1 and 6 days after surgery. Recovery will be assessed 3 times a day (7.00 am, 12.00 am, 6.00 pm)

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien Venara, MD, Principal Investigator — University Hospital Center of Angers
Locations (1):
- University Hospital Center, Angers, France

IPD SHARING:
Plan to Share IPD: No